CLINICAL TRIAL: NCT05063214
Title: Muscle Evaluation of Patients Infected by the Coronavirus Requiring Mechanical Ventilation
Brief Title: Muscle Evaluation of Patients Infected by the Coronavirus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Other Study IDs: 49075421.0.0000.0071; 4.923.576 (Other: Hospital Israelita Albert Einstein Ethics Committee)
Record Dates: First submitted 2021-09-04; First posted 2021-10-01 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: SARS-CoV-2 Acute Respiratory Disease
Keywords: Coronavirus; SARS-CoV-2; COVID-19; Intensive Care Units; Ultrasonography
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ultrasound assessment: Muscle ultrasound evaluation
  Interventions: Diagnostic Test: Muscle ultrasound evaluation

INTERVENTIONS:
Diagnostic Test: Muscle ultrasound evaluation — Muscle ultrasound evaluation will be performed in patients admitted with COVID-19 requiring invasive mechanical ventilation. The measurements of thickness and thickening fraction will occur for diaphragm, abdominal - rectus abdominis, internal oblique, external oblique and transverse abdomen - and parasternal intercostal muscles. Serial measurements of the thickness and echogenicity of the quadriceps femoris muscle will also be performed.

SUMMARY:
Patients with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) presents risk to develop muscle weakness associated with prolonged period of mechanical ventilation support and hospital stay.

DETAILED DESCRIPTION:
Intensive care unit (ICU) acquired muscle weakness affects both respiratory and peripheral muscles and can contribute to worsen clinical and functional outcomes. In this way, ultrasonography muscle evaluation could help to identify early alterations guiding the therapeutic planning and allowing to monitor the interventions performed. Therefore, the investigators intend to follow up mechanically ventilated patients with confirmed diagnosis of COVID-19 during ICU stay to quantify the diaphragm, parasternal intercostal, abdominals and femoral quadriceps muscles thickness assessed by ultrasonography. Additionally, functional capacity, frailty and level of physical activity will be evaluated and followed for pre-admission condition and 30, 90 and 180 days after hospital discharge .

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to ICU
* having a confirmed diagnosis of COVID-19
* requiring invasive mechanical ventilation.

Exclusion Criteria:

* exclusive palliative care;
* neuromuscular diseases;
* patients who evolve with the need for lower limb amputation;
* previous known diaphragm malformations and dysfunctions;
* patients transferred from other institutions under invasive mechanical ventilation;
* clinical conditions that make the respiratory and peripheral muscle assessment through ultrasound unfeasible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SARS-CoV-2 patients admitted to the intensive care unit requiring invasive mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Muscle thickness | Day 1, 5, and within 24 hours after ICU discharge.
  Change in the thickness of the diaphragm and quadriceps femoris muscles.

SECONDARY OUTCOMES:
Respiratory muscle thickness | At the end of data collection, within 24 hours after ICU discharge.
  Change in the thickness of the intercostal and abdominal wall muscles.
Muscle thickness and functional outcomes | At the end of data collection, within 24 hours after ICU discharge.
  Verify the correlation between quadriceps femoris muscle thickness change and echogenicity with functional outcomes (Barthe Index, International Physical Activities Questionnaire, and the Clinical Frailty Score).
Grip strength and clinical outcomes | At the end of data collection, within 24 hours after ICU discharge.
  Verify the correlation between grip strength (measured by the Dynamometer Grip Strength) and clinical outcomes (Barthe Index, International Physical Activities Questionnaire, and the Clinical Frailty Score).
Mobility level correlation with clinical and functional outcomes | At the end of data collection, within 24 hours after ICU discharge.
  Verify the correlation between mobility level (measured by the Perme Intensive Care Unit Mobility Score) with clinical and functional outcomes (Barthe Index, International Physical Activities Questionnaire, and the Clinical Frailty Score).

CONTACTS AND LOCATIONS:
Overall Officials: Caroline G Mól, PT, Study Chair — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) collected during the study that underlie results reported will be shared after de-identification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available at the end of the study, as soon as the manuscript became published in a journal (following publication). No end date (data will be available indefinitely).
Access Criteria: Researchers who provide a methodologically sound proposal and/or investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.

REFERENCES:
- [Background] Vanhorebeek I, Latronico N, Van den Berghe G. ICU-acquired weakness. Intensive Care Med. 2020 Apr;46(4):637-653. doi: 10.1007/s00134-020-05944-4. Epub 2020 Feb 19. PMID 32076765
- [Background] Conway H, Lau G, Zochios V. Personalizing Invasive Mechanical Ventilation Strategies in Coronavirus Disease 2019 (COVID-19)-Associated Lung Injury: The Utility of Lung Ultrasound. J Cardiothorac Vasc Anesth. 2020 Oct;34(10):2571-2574. doi: 10.1053/j.jvca.2020.04.062. Epub 2020 May 15. No abstract available. PMID 32425463
- [Background] Patel Z, Franz CK, Bharat A, Walter JM, Wolfe LF, Koralnik IJ, Deshmukh S. Diaphragm and Phrenic Nerve Ultrasound in COVID-19 Patients and Beyond: Imaging Technique, Findings, and Clinical Applications. J Ultrasound Med. 2022 Feb;41(2):285-299. doi: 10.1002/jum.15706. Epub 2021 Mar 27. PMID 33772850
- [Background] Shi Z, de Vries HJ, Vlaar APJ, van der Hoeven J, Boon RA, Heunks LMA, Ottenheijm CAC; Dutch COVID-19 Diaphragm Investigators. Diaphragm Pathology in Critically Ill Patients With COVID-19 and Postmortem Findings From 3 Medical Centers. JAMA Intern Med. 2021 Jan 1;181(1):122-124. doi: 10.1001/jamainternmed.2020.6278. PMID 33196760
- [Background] Vivier E, Mekontso Dessap A, Dimassi S, Vargas F, Lyazidi A, Thille AW, Brochard L. Diaphragm ultrasonography to estimate the work of breathing during non-invasive ventilation. Intensive Care Med. 2012 May;38(5):796-803. doi: 10.1007/s00134-012-2547-7. Epub 2012 Apr 5. PMID 22476448
- [Background] Goligher EC, Fan E, Herridge MS, Murray A, Vorona S, Brace D, Rittayamai N, Lanys A, Tomlinson G, Singh JM, Bolz SS, Rubenfeld GD, Kavanagh BP, Brochard LJ, Ferguson ND. Evolution of Diaphragm Thickness during Mechanical Ventilation. Impact of Inspiratory Effort. Am J Respir Crit Care Med. 2015 Nov 1;192(9):1080-8. doi: 10.1164/rccm.201503-0620OC. PMID 26167730
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Sklar MC, Dres M, Fan E, Rubenfeld GD, Scales DC, Herridge MS, Rittayamai N, Harhay MO, Reid WD, Tomlinson G, Rozenberg D, McClelland W, Riegler S, Slutsky AS, Brochard L, Ferguson ND, Goligher EC. Association of Low Baseline Diaphragm Muscle Mass With Prolonged Mechanical Ventilation and Mortality Among Critically Ill Adults. JAMA Netw Open. 2020 Feb 5;3(2):e1921520. doi: 10.1001/jamanetworkopen.2019.21520. PMID 32074293
- [Background] Itagaki T, Nakanishi N, Takashima T, Ueno Y, Tane N, Tsunano Y, Nunomura T, Oto J. Effect of controlled ventilation during assist-control ventilation on diaphragm thickness : a post hoc analysis of an observational study. J Med Invest. 2020;67(3.4):332-337. doi: 10.2152/jmi.67.332. PMID 33148911
- [Background] Goligher EC, Dres M, Fan E, Rubenfeld GD, Scales DC, Herridge MS, Vorona S, Sklar MC, Rittayamai N, Lanys A, Murray A, Brace D, Urrea C, Reid WD, Tomlinson G, Slutsky AS, Kavanagh BP, Brochard LJ, Ferguson ND. Mechanical Ventilation-induced Diaphragm Atrophy Strongly Impacts Clinical Outcomes. Am J Respir Crit Care Med. 2018 Jan 15;197(2):204-213. doi: 10.1164/rccm.201703-0536OC. PMID 28930478
- [Background] Goligher EC, Laghi F, Detsky ME, Farias P, Murray A, Brace D, Brochard LJ, Bolz SS, Rubenfeld GD, Kavanagh BP, Ferguson ND. Measuring diaphragm thickness with ultrasound in mechanically ventilated patients: feasibility, reproducibility and validity. Intensive Care Med. 2015 Apr;41(4):642-9. doi: 10.1007/s00134-015-3687-3. Epub 2015 Feb 19. PMID 25693448
- [Background] Vivier E, Roussey A, Doroszewski F, Rosselli S, Pommier C, Carteaux G, Mekontso Dessap A. Atrophy of Diaphragm and Pectoral Muscles in Critically Ill Patients. Anesthesiology. 2019 Sep;131(3):569-579. doi: 10.1097/ALN.0000000000002737. PMID 31094757
- [Background] Parry SM, El-Ansary D, Cartwright MS, Sarwal A, Berney S, Koopman R, Annoni R, Puthucheary Z, Gordon IR, Morris PE, Denehy L. Ultrasonography in the intensive care setting can be used to detect changes in the quality and quantity of muscle and is related to muscle strength and function. J Crit Care. 2015 Oct;30(5):1151.e9-14. doi: 10.1016/j.jcrc.2015.05.024. Epub 2015 Jun 3. PMID 26211979
- [Background] Nakanishi N, Oto J, Ueno Y, Nakataki E, Itagaki T, Nishimura M. Change in diaphragm and intercostal muscle thickness in mechanically ventilated patients: a prospective observational ultrasonography study. J Intensive Care. 2019 Dec 2;7:56. doi: 10.1186/s40560-019-0410-4. eCollection 2019. PMID 31827804
- [Background] Zambon M, Beccaria P, Matsuno J, Gemma M, Frati E, Colombo S, Cabrini L, Landoni G, Zangrillo A. Mechanical Ventilation and Diaphragmatic Atrophy in Critically Ill Patients: An Ultrasound Study. Crit Care Med. 2016 Jul;44(7):1347-52. doi: 10.1097/CCM.0000000000001657. PMID 26992064
- [Background] Matamis D, Soilemezi E, Tsagourias M, Akoumianaki E, Dimassi S, Boroli F, Richard JC, Brochard L. Sonographic evaluation of the diaphragm in critically ill patients. Technique and clinical applications. Intensive Care Med. 2013 May;39(5):801-10. doi: 10.1007/s00134-013-2823-1. Epub 2013 Jan 24. PMID 23344830
- [Background] Tuinman PR, Jonkman AH, Dres M, Shi ZH, Goligher EC, Goffi A, de Korte C, Demoule A, Heunks L. Respiratory muscle ultrasonography: methodology, basic and advanced principles and clinical applications in ICU and ED patients-a narrative review. Intensive Care Med. 2020 Apr;46(4):594-605. doi: 10.1007/s00134-019-05892-8. Epub 2020 Jan 14. PMID 31938825
- [Background] Formenti P, Umbrello M, Dres M, Chiumello D. Ultrasonographic assessment of parasternal intercostal muscles during mechanical ventilation. Ann Intensive Care. 2020 Sep 7;10(1):120. doi: 10.1186/s13613-020-00735-y. PMID 32894372
- [Background] Shi ZH, de Vries H, de Grooth HJ, Jonkman AH, Zhang Y, Haaksma M, van de Ven PM, de Man AAME, Girbes A, Tuinman PR, Zhou JX, Ottenheijm C, Heunks L. Changes in Respiratory Muscle Thickness during Mechanical Ventilation: Focus on Expiratory Muscles. Anesthesiology. 2021 May 1;134(5):748-759. doi: 10.1097/ALN.0000000000003736. PMID 33711154
- [Background] Tillquist M, Kutsogiannis DJ, Wischmeyer PE, Kummerlen C, Leung R, Stollery D, Karvellas CJ, Preiser JC, Bird N, Kozar R, Heyland DK. Bedside ultrasound is a practical and reliable measurement tool for assessing quadriceps muscle layer thickness. JPEN J Parenter Enteral Nutr. 2014 Sep;38(7):886-90. doi: 10.1177/0148607113501327. Epub 2013 Aug 26. PMID 23980134